CLINICAL TRIAL: NCT01745887
Title: A Multi-Center, Double Masked, Randomized, Placebo-Controlled, Dose-Ranging Study of EBI-005 Ophthalmic Solution Versus Placebo in Subjects With Dry Eye Syndrome
Brief Title: A Multi-Center Study Subjects With Dry Eye Syndrome
Acronym: EBI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eleven Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBI-005-2
Record Dates: First submitted 2012-12-04; First posted 2012-12-10 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Dry Eye Syndrome
Keywords: Dry Eye Syndrome; Interleukin 1 Receptor Inhibitor
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- EBI-005-2 5mg/ml (Active Comparator): Administration: 3 times per day
  Interventions: Drug: EBI-005-2
- EBI-005-2 20 mg/ml (Active Comparator): Administration: 3 times per day
  Interventions: Drug: EBI-005-2
- EBI-005-2 Placebo (Placebo Comparator): Administration: 3 times per day

INTERVENTIONS:
Drug: EBI-005-2 — The investigational drug EBI-005-2, is an intervention to three different study arms. One arm gets 5mg/ml, the other gets 20mg/ml and the last arm is Placebo.
  Arms: EBI-005-2 20 mg/ml; EBI-005-2 5mg/ml

SUMMARY:
This is a Phase 1b, multi-center, double-masked, randomized, placebo-controlled, parallel-group study designed to evaluate the safety and biological activity of two doses of EBI-005 ophthalmic solution versus placebo in subjects with moderate to severe Dry Eye Syndrome. Approximately 72 subjects will be enrolled and randomized in this study at up to 9 centers located in the United States (US). Subjects will be enrolled in two groups or cohorts. The first enrollment group will consist of 33 subjects.

DETAILED DESCRIPTION:
* To investigate the safety and tolerability of EBI-005 ophthalmic solution compared to placebo in the treatment of patients with moderate to severe Dry Eye Syndrome (DES).
* To evaluate pharmacokinetic (PK) parameters and immunogenicity of two different doses of EBI-005 ophthalmic solution.
* To investigate the biological activity of multiple doses of EBI-005 ophthalmic solution compared to placebo as assessed by both objective and subjective assessments.
* To investigate the comparative dose response of two different doses of EBI-005 ophthalmic solution.
* To investigate the comparative tolerability of two different doses of EBI-005 ophthalmic solution.
* To identify key biomarkers in the diagnosis and management of subjects with DES.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to any study related procedures
* Are 18 years of age or older
* Are women of child bearing potential (WOCBP) who are non-pregnant, non-lactating and sexually inactive (abstinent) for 14 days prior to Visit 1
* Are willing and able to follow instructions and can be present for the required study visits for the duration of the study
* Have a history of Dry Eye Syndrome in both eyes supported by a previous clinical diagnosis
* Have ongoing Dry Eye Syndrome, in the same eye or both eyes, as defined by the following criteria:

  1. A score of ≥23 on OSDI
  2. A corneal fluorescein staining score of ≥6 (NEI scale)
* Have normal lid anatomy
* Are willing to withhold artificial tears for the duration of the study, with the exception of the study provided artificial tears: Refresh Plus®.

Exclusion Criteria: Subjects may not:

* Have previously used an IL-1 blocker (e.g., Anakinra, Rilonacept or Ilaris).
* Have an OSDI score ≥90
* Have a corneal fluorescein staining score of 15 (NEI scale). NOTE: If one of two eyes has a corneal fluorescein staining score of 15, the subject may be eligible.
* Within 30 days prior to the screening visit (Visit 1) have taken: Topical cyclosporine (Restasis®) Ocular corticosteroids Autologous serum Topical ocular antibiotics Topical ocular antihistamines or mast cell stabilizers Topical or nasal vasoconstrictors
* Within 30 days prior to the screening visit (Visit 1) have altered the dose of tetracycline compounds (tetracycline, doxycycline or minocycline).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
OSDI (Ocular Surface Disease Index) | 2 months
  OSDI is a subject assessment tool to determine subject Dry Eye Syndrome symptoms

SECONDARY OUTCOMES:
Change from baseline in total corneal fluorescein staining | 2 months
  Corneal staining assessment will be performed using methods developed by the NEI Dry Eye Workshop.
Symptom Assessment in Dry Eye (Modified SANDE) | 2 months
  Patient Reported Outcome using a Visual Analog Scale for Modified SANDE.

OTHER OUTCOMES:
Gene transcription levels measured from cells collected via impression cytology | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Goldstein, MD, Study Director — Eleven Biotherapeutics
Locations (8):
- United States (8):
  - Investigational Site, Artesia, California
  - Investigational Site, Ranchero Cordova, California
  - Investigational Site, Torrence, California
  - Investigational Site, Kansas City, Missouri
  - Investigational Site, Washington, Missouri
  - Investigational Site, Cleveland, Ohio
  - Investigational Site, San Antonio, Texas
  - Investigational Site, Norfolk, Virginia